CLINICAL TRIAL: NCT06155851
Title: Prevalence of Hiatus Hernia in Gastro-Esophageal Reflux Disease Patients Underwent Upper Endoscopy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Ibrahim Aboelela, resident doctor, Assiut University
Other Study IDs: Prevalence of Hiatus Hernia in
Record Dates: First submitted 2023-09-11; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Hiatus Hernia
MeSH Terms: conditions — Hernia, Hiatal | interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Upper Endoscopy — Endescopy

SUMMARY:
To study the prevalence of hiatus hernia in GERD patients underwent upper endoscopy To study the effect of hiatus hernia on the severity of GERD symptoms.

DETAILED DESCRIPTION:
Gastro-esophageal reflux disease (GERD) is a common problem for which patients seek care from a broad array of primary care providers, medical sub-specialists, and surgeons.

It is estimated that 10 to 20 percent of people in Western countries have GERD, when defined as heartburn or regurgitation at least once a week. (Chapelle, et al. 2021)

The practice guidelines for GERD recommend diagnostic testing in the presence of alarm symptoms, which include dysphagia, odynophagia, weight loss, gastrointestinal bleeding, and anemia.

A detailed history of the pattern, severity, and duration of alarm symptoms is essential. (Katz, et al., 2022) Hiatus hernia refers to condition in which elements of the abdominal cavity, most commonly the stomach, herniate through the esophageal hiatus into the mediastinum.

Hiatus hernia is a frequent finding during upper gastrointestinal endoscopy. Type I hiatal hernia is the sliding hiatal hernia, which accounts for more than 95% of all hiatal hernias with the remaining 5% being Para-esophageal hiatus hernias (Kotekar, et al 2021)

Endoscopy is a common diagnostic tool in the evaluation of patients with upper gastrointestinal pathology, specifically gastroesophageal reflux disease (GERD) and hiatal hernia.

The relationship between these two disease processes are relatively intertwined and have clinical significance given the fact patients with hiatal hernia may be more likely to have acid reflux and there is a close relationship with hiatal hernia size and incidence of reflux disease. (Gomaa, et al 2022) Worldwide, it is believed that the relation between hiatus hernia and gastro-esophageal reflux disease (GERD) have varied considerably.

In our locality the prevalence of hiatal hernia in GERD patients and the effect of hiatal hernia on the severity of GERD symptoms is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older, Patients with GERD symptoms who don't respond to PPI therapy (8 weeks ) or cases with alarm symptoms (dysphagia, anemia ,vomiting , weight loss , GI bleeding , onset of symptoms in old age ,..etc)

Exclusion Criteria:

* Complete PPI responder. Patient with any contraindication for endoscopy . Refusal of participation

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all cases matching inclusion criteria during the time of the study will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
To study the prevalence of hiatus hernia in GERD patients underwent upper endoscopy To study the effect of hiatus hernia on the severity of GERD symptoms. | prospective cohort syudy_ up to 1 year
  To study the prevalence of hiatus hernia in GERD patients underwent upper endoscopy To study the effect of hiatus hernia on the severity of GERD symptoms.

REFERENCES:
- [Background] Levin JG, Seidman JG. Selective packaging of host tRNA's by murine leukemia virus particles does not require genomic RNA. J Virol. 1979 Jan;29(1):328-35. doi: 10.1128/JVI.29.1.328-335.1979. PMID 219227
- [Background] Daraz B, Piela A. [Treatment and prevention of EPH-gestosis]. Pieleg Polozna. 1978;(5):7-8. No abstract available. Polish. PMID 254272
- [Background] Kromer W, Freundt KJ. [In vitro inhibition of oxidative N-demethylation with carbon disulfide]. Arzneimittelforschung. 1976 Feb;26(2):189-94. German. PMID 7280
- [Background] Newton JM, Razzo RN. Proceedings: The influence of formulation variables on the in vitro release of drug from hard gelatin capsules. J Pharm Pharmacol. 1975 Dec;27 Suppl?-2:79P. No abstract available. PMID 2756
- [Background] Herold G, Stephan B, Menzel T. [The behavior of bioelements during long-term parenteral feeding]. Infusionsther Klin Ernahr. 1979 Apr;6(2):105-10. German. PMID 107121